CLINICAL TRIAL: NCT06576076
Title: Characterizing Proximal Risk for Depressive Symptoms and Suicidal Ideation With Acute Cannabis Use and Withdrawal Among Adolescents Using Ecological Momentary Assessment
Brief Title: Cannabis, Linked Emotions, and Adolescent Risk Study
Acronym: CLEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Randi Melissa Schuster, Associate Professor; Director of School-Based Research and Program Development, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024P002417; 1R01DA054145-01A1 (NIH)
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use; Depression; Suicidal Ideation; Adolescent Behavior
MeSH Terms: conditions — Depression; Suicidal Ideation; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Following a shared two-week baseline assessment period (Arm 1) for all enrolled participants, participants will be split into 2 arms, randomly assigned to one of two interventions (Arms 2 or 3, CB-Abst or CB-Mon).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cannabis Abstinence (CB-Abst) (Experimental): Those randomized to the abstinence condition will be asked to stop using cannabis for eight weeks. They will participate in a contingency management protocol, which uses an escalating remuneration schedule to incentivize abstinence. Abstinence is confirmed biochemically via progressively decreasing values of creatinine-adjusted THCCOOH.
  Interventions: Behavioral: Contingency management for cannabis abstinence
- Cannabis Monitoring (CB-Mon) (No Intervention): Those randomized to the monitoring condition will be asked to make no changes to their cannabis use frequency or dose for the duration of the eight week study.
- Pre-intervention Pooled Groups (EMA Phase 1 Only) (No Intervention): All enrolled participants will participate in approximately two weeks of EMA data collection prior to being randomized and starting intervention procedures to characterize mood during baseline use as usual (CB-Abst or CB-Mon).

INTERVENTIONS:
Behavioral: Contingency management for cannabis abstinence — Those randomized to the abstinence condition (CB-Abst) will be incentivized using an escalating reinforcement schedule for eight weeks of cannabis abstinence.
  Arms: Cannabis Abstinence (CB-Abst)

SUMMARY:
The goal of this study is to disentangle relationships between acute cannabis use and withdrawal on proximal depression and suicide risk and recovery in adolescents ages 12-18 years by incorporating time-varying patterns of substance use, mood, and SI. This project aims to guide the development of scalable, individualized, accessible, and affordable interventions aimed to reduce depression and suicide risk among adolescents.

DETAILED DESCRIPTION:
We will recruit 200 community-based adolescents, ages 12-18 years, with daily or near daily cannabis use and current depression symptoms. Participants will be enrolled in a 10-week, 3-phased, mixed-methods protocol. All participants will complete a 2 week baseline phase (Phase 1) involving real-time, ambulatory smartphone monitoring (ecological momentary assessment; EMA) during which they will use cannabis per usual to quantify the temporal relationship between use and mood and SI, and the within- (e.g., concurrent other substance use, social context of use) and between-subject factors (e.g., severity of cannabis use, depression and SI) that moderate these linkages. We will work with participants schedule to ensure that the start of this 2-week baseline phase coincides with when they do not anticipate any major deviations from their typical pattern of cannabis use (e.g., family vacation, exam week). After the baseline phase, participants will be scheduled for the randomization component of the study, which will employ a 2-arm, within-subject, parallel group design to examine the effects of short- and longer-term cannabis withdrawal across 8 weeks of cannabis abstinence on depression and SI. Participants will be randomized to 8 weeks of abstinence with contingency management (CB-Abst; n=100) or non-contingent monitoring with no abstinence requirement (CBMon; n=100). Randomization will occur in a 1:1 ratio in blocks of 6 based on a computerized scheme developed by the study statistician. Randomization will be stratified by age, sex, and depression severity. A key aspect of the approach is that the 8-week period is long enough to observe true changes due to cannabis discontinuation, separate from effects of cannabis withdrawal, and residual cannabinoid exposure. Both groups will complete 1-week of EMA in weeks 1 (Phase 2) and 8 (Phase 3) of the randomized study period. In addition to the 3 waves of smartphone, EMA data collection, participants will complete 12 study visits across ~10 weeks. Visits will entail collection of urine samples for verification of self-reported use and abstinence verification (for CB-Abst during the randomization phase), as well as brief questionnaires and interviews on interim substance use, craving, withdrawal, mood symptoms, and SI.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-18;
* Current daily or near daily cannabis use (i.e., use ≥ 4 days per week on average; Timeline Followback);
* Score ≥ 5 on PHQ-9;
* Access to an internet-capable smartphone (iOS or Android);
* Provision of at least 1 collateral contact for risk monitoring;
* Provision of informed assent (or consent if 18 years or older) and parent/guardian consent if <age 18;
* Greater than 50% response rate to EMA prompts during the first EMA phase;
* No immediate plan to discontinue cannabis use in the next 3 months;
* Positive toxicology result for cannabis on baseline urinalysis.

Exclusion Criteria:

* Any factor that impairs ability to comprehend and effectively participate, including acute intoxication at time of consent;
* Cannabis use >4 times/day on average (to maximize likelihood of capturing mood and SI during non-use times);
* Inability to speak/write English fluently;
* Gross cognitive impairment, for example due to florid psychosis, intellectual disability, developmental delay, or neurodegenerative disease;
* Current epilepsy diagnosis;
* Individuals who are under the legal protection of the government or state (wards of the state);
* Response of "No" to the knowledge check question regarding EMA suicidality response time;
* Inability to wear Fitbit device.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Cannabis use in the last hour | Weeks 1 - 2 (EMA Phase 1; Baseline Use as Usual)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a binary rating as to whether cannabis was used in the last hour, either 0 (No use) or 1 (Use in the last hour). We will examine data from all participants prior to randomization to experimental arms (Pre-intervention Pooled Groups arm).
Aim 1: Motivation to use cannabis to improve mood collected | Weeks 1 - 2 (EMA Phase 1; Baseline Use as Usual)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. We will use the subset of responses following cannabis use in the last hour. The outcome is a rating for whether cannabis was used to improve negative mood, from 1 (No, not at all) to 100 (Yes, very much). Higher ratings indicate greater motivation to use cannabis to improve negative mood. We will examine data from all participants prior to randomization to experimental arms (Pre-intervention Pooled Groups arm).
Aim 2: Depleted mood | Weeks 1 - 3, Week 10 (EMA Phase 2-3; Randomized Withdrawal then Sustained Abstinence)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a composite score of depleted mood computed as the average over 5 ratings each assessed on a 0 (No, not at all) - 100 (Yes, very much) scale with the following question prompt: Right now how much do you feel [MOOD] (sub in Sad/Self-hatred/Numb/Hopeless/Fatigued). Higher ratings indicate worse feelings of depleted mood. We will examine data for participants split between the two experimental arms (CB-Abst versus CB-Mon).
Aim 2: Negative cognitive impact | Weeks 1 - 3, Week 10 (EMA Phase 2-3; Randomized Withdrawal then Sustained Abstinence)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a composite score of negative cognitive impact computed as the average over 2 ratings each assessed on a 0 (No, not at all) - 100 (Yes, very much) scale with the following question prompt: Right now how much do you feel [MOOD] (sub in Disinterested/Inattentive). Higher ratings indicate worse feelings of negative cognitive impact. We will examine data for participants split between the two experimental arms (CB-Abst versus CB-Mon).
Aim 2: Negative activation | Weeks 1 - 3, Week 10 (EMA Phase 2-3; Randomized Withdrawal then Sustained Abstinence)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a composite score of negative activation computed as the average over 3 ratings each assessed on a 0 (No, not at all) - 100 (Yes, very much) scale with the following question prompt: Right now how much do you feel [MOOD] (sub in Agitated/Irritated/Anxious). Higher ratings indicate worse feelings of negative activation. We will examine data for participants split between the two experimental arms (CB-Abst versus CB-Mon).
Aim 2: Passive suicidal ideation | Weeks 1 - 3, Week 10 (EMA Phase 2-3; Randomized Withdrawal then Sustained Abstinence)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a composite score of passive suicidal ideation computed as the average over 3 ratings each assessed on a 0 (No, not at all) - 100 (Yes, very much) scale with the following question prompt: Right now how strong is your [IDEATION] (sub in Thoughts about death/Wishing suffering could be over/Better off as dead). Higher ratings indicate worse passive suicidal ideation. We will examine data for participants split between the two experimental arms (CB-Abst versus CB-Mon).
Aim 2: Suicidal urges | Weeks 1 - 3, Week 10 (EMA Phase 2-3; Randomized Withdrawal then Sustained Abstinence)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a rating to the following prompt: right now how strong is your intention to kill yourself, from 0 (No, not at all) to 100 (Yes, very much). Higher ratings indicate worse suicidal urges. We will examine data for participants split between the two experimental arms (CB-Abst versus CB-Mon).
Aim 2: Non-suicidal self-injury urges | Weeks 1 - 3, Week 10 (EMA Phase 2-3; Randomized Withdrawal then Sustained Abstinence)
  Responses will be collected via ecological momentary assessment based on 7-9 random prompts a day. The outcome is a rating to the following prompt: right now how strong is your desire to hurt your body, from 0 (No, not at all) to 100 (Yes, very much). Higher ratings indicate worse self-injury urges. We will examine data for participants split between the two experimental arms (CB-Abst versus CB-Mon).

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hopsital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
As outlined in the approved Data Management and Sharing Plan, IPD will be deposited in the NIMH Data Archive. This is a free data repository open to qualified researchers from all mental health and other research communities to share, archive, cite, access, and explore research data. Clinical data necessary to validate and replicate research findings, including questionnaires, interviews, ecological momentary assessment data, urine drug test results, and Fitbit recordings, will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Scientific data will be available one year after the grant end date specified on the first Notice of Award. Scientific data included in published manuscripts will be made available at the time of publication. Scientific data and the code/software/tools used to development the published or submitted dataset will be shared at the time of data submission or publication and maintained for no shorter than five years.
Access Criteria: Data access will be controlled. In order to access shared data, qualified researchers will be required to complete a data use certification and receive approval from NDA Data Access Committee.

REFERENCES:
- [Derived] Feibus I, Mahiques MB, Costello M, Potter K, Bentley KH, Hoeppner BB, Liu L, Evohr B, Yan L, Gilman J, Evins AE, Kossowsky J, Schuster RM. Characterizing proximal risk for depressive symptoms and suicidal ideation with acute cannabis use and withdrawal among adolescents using ecological momentary assessment: Study protocol. PLoS One. 2025 Dec 18;20(12):e0338790. doi: 10.1371/journal.pone.0338790. eCollection 2025. PMID 41411314